CLINICAL TRIAL: NCT06019156
Title: Effectiveness of Metaverse Space-based Exercise Video Distribution in Young Adults: A Randomized Controlled Trial
Brief Title: Effectiveness of Metaverse Space-based Exercise Video Distribution in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hiroshima University (Other)
Responsible Party: Principal Investigator, Rami Mizuta, Principal Investigator, Doctoral student of Graduate School of Biomedical and Health Sciences Hiroshima University, Hiroshima University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: C2022-0044
Record Dates: First submitted 2023-08-06; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- metaverse group (Experimental)
  Interventions: Behavioral: Exercise video distribution of Metaverse
- YouTube group (Active Comparator)
  Interventions: Behavioral: Exercise video distribution of YouTube
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Exercise video distribution of Metaverse — Participants received a 10-minute exercise video each week with a load of about 4 to 8 metabolic equivalents of task (METs) in the metaverse space, for eight videos delivered to encourage exercise.
  Arms: metaverse group
Behavioral: Exercise video distribution of YouTube — Participants view exercise videos with the same content as the metaverse group.
  Arms: YouTube group

SUMMARY:
This study explored whether exercise video distribution using metaverse space is effective in increasing physical activity among young people, along with mental health and locomotive function. This is a randomized parallel-group study. Participants will be assigned to 3 groups: a metaverse group, a YouTube group, and a control group. The metaverse group will receive eight 10-minute exercise videos each week with approximately 4 to 8 METs (metabolic equivalents of task) in the metaverse space to encourage exercise, and the YouTube group will receive access to the same exercise videos as the metaverse group. The control group was given no specific instructions.

The intervention period was 8 weeks, and physical activity and other items were measured before and after the intervention. These pre- and post-intervention measurements will be used to determine whether the delivery of exercise videos via Metaverse is effective in increasing physical activity in young adults.

ELIGIBILITY:
Inclusion Criteria:

* individuals aged 18-30 at the time of obtaining consent
* who owned a smartphone or computer and had internet access
* who did not belong to an exercise community, such as a sports club

Exclusion Criteria:

* individuals who had a history of a disease that prohibited exercise
* individuals whose physical activity was > 3000 metabolic equivalents of task (METs)/week
* pregnant (or possibly pregnant) women

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2022-12-11 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Physical activity | The pre-measurement answered the most recent week, and the post-measurement responded to the next week after the 8 weeks intervention was finished.
  The short form of the International Physical Activity Questionnaire Short Form was used to measure the effect of an intervention.

SECONDARY OUTCOMES:
Well-being | Pre- and post- 8 weeks intervention
  The Japanese version of the World Health Organization Five-Well-Being Index was used.
Psychological distress | Pre- and post- 8 weeks intervention
  The 6-item Kessler Scale as a nonspecific psychological distress scale was used.
Locomotive syndrome risk tests | Pre- and post- 8 weeks intervention
  We used the 25-question geriatric locomotive function scale.
Social capital | Pre- and post- 8 weeks intervention
  The social capital questions consisted of 11 items related to civic participation, social cohesion, and reciprocity, with a perfect score of 11 and higher scores indicating stronger social connections.
Quality of life (QOL) | Pre- and post- 8 weeks intervention
  The Japanese version of the 26-item World Health Organization QOL measure was used to assess QOL.

CONTACTS AND LOCATIONS:
Overall Officials: Yukio Urabe, PhD, Principal Investigator — Hiroshima University
Locations (1):
- Hiroshima University, Hiroshima, Japan

IPD SHARING:
Plan to Share IPD: No
There are no plans to make Individual Participant Data (IPD) available to other researchers.

REFERENCES:
- [Derived] Mizuta R, Maeda N, Tashiro T, Suzuki Y, Kuroda S, Ishida A, Oda S, Watanabe T, Tamura Y, Komiya M, Urabe Y. Effectiveness of Metaverse Space-Based Exercise Video Distribution in Young Adults: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2024 Jan 16;12:e46397. doi: 10.2196/46397. PMID 38227355